CLINICAL TRIAL: NCT03444558
Title: Effect of a Natural Supplement Containing Chlorogenic Acid and Luteolin on Cardio-metabolic Risk Factors in Patients With Metabolic Syndrome
Brief Title: Effects of Natural Supplement Containing Chlorogenic Acid and Luteolin on Cardio-metabolic Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Collaborators: University of Catania (Other)
Responsible Party: Principal Investigator, Manfredi Rizzo, MD, PhD, Associate Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Natural Supplement
Record Dates: First submitted 2017-06-05; First posted 2018-02-23 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Metabolic Syndrome
Keywords: metabolic parameters; cardio-metabolic parameters
MeSH Terms: conditions — Metabolic Syndrome | interventions — Luteolin

STUDY DESIGN:
Intervention Model Description: placebo-controlled study
Who Masked: Participant, Investigator
Masking Description: double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Supplement (Experimental): 50 subjects with the metabolic syndrome receiving natural supplement containing chlorogenic acid and luteolin (450 mg/die)
  Interventions: Dietary Supplement: Natural supplement containing chlorogenic acid and luteolin
- Placebo (Placebo Comparator): 50 subjects with the metabolic syndrome receiving placebo (without any active ingredients)
  Interventions: Other: Placebo (without any active ingredients)

INTERVENTIONS:
Dietary Supplement: Natural supplement containing chlorogenic acid and luteolin — 50 eligible subjects will receive natural supplement as the oral pills at a fixed dose of 1 pill/day (450 mg/day) for 6 months, as add-on therapy to the ongoing treatment, maintained at fixed doses for the entire study.
  Arms: Dietary Supplement
Other: Placebo (without any active ingredients) — 50 eligible subjects will receive placebo (without any active ingredients) at a fixed dose of 1 pill/day for 6 months, as add-on therapy to the ongoing treatment, maintained at fixed doses for the entire study.
  Arms: Placebo

SUMMARY:
Clinical trial about beneficial effects of natural ingredient containing chlorogenic acid and luteolin on liver health and conditions related to liver (such as metabolic syndrome) for general body health.

DETAILED DESCRIPTION:
This is one randomized, double-blind, placebo-controlled study. The purpose of the present study is to evaluate and/or elucidate the role of the natural supplement, containing chlorogenic acid (10-12%) and luteinyl-7-glucoside (2-4%), on cardio-metabolic risk factors.

The research hypothesis is to evaluate whether natural supplement containing chlorogenic acid and luteolin (Puraltilix, BIONAP SRL, Catania, Italy) may improve several cardio-metabolic parameters in subjects with the metabolic syndrome.

All subjects will be evaluated at baseline and after 6 months of treatment (with natural supplement or placebo).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged >18 years with the metabolic syndrome (as defined by the international criteria: Alberti KG, et al. Circulation. 2009; 120: 1640-5);
* BMI> 25 kg/m^2;
* Subjects able to swallow whole tablets;
* Informed consent obtained prior to any study-related activities.

Exclusion Criteria:

* Pregnancy or willingness to become pregnant;
* Severe liver dysfunction (ALT >2.5 times upper limit of normal);
* Severe renal failure (eGFR<60 mL/min/1.73 m2 using the MDRD formula);
* Severe infections at the discretion of the investigator (such as HIV, HBV and HCV);
* History or presence of malignant neoplasms within the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Effect of natural supplement on metabolic parameters including body weight and Body Mass Index (BMI) | Change from baseline to 6 months of the supplementation
  Effect of natural supplement containing chlorogenic acid and luteolin on metabolic parameters, including body weight (kg) and height (m) that will be combined to report BMI in kg/m^2.
Effect of natural supplement on metabolic parameters including waist circumference | Change from baseline to 6 months of the supplementation
  Effect of natural supplement containing chlorogenic acid and luteolin on metabolic parameters, including waist circumference (cm).
Effect of natural supplement on metabolic parameters including plasma lipids | Change from baseline to 6 months of the supplementation
  Effect of natural supplement containing chlorogenic acid and luteolin on metabolic parameters, including plasma lipids (total cholesterol, triglycerides, high-density lipoprotein cholesterol HDL-C) (mmol/l), while low-density lipoprotein cholesterol (LDL-C) will be calculated using the Friedewald formula.
Effect of natural supplement on metabolic parameters including glucose metabolism parameters | Change from baseline to 6 months of the supplementation
  Effect of natural supplement containing chlorogenic acid and luteolin on metabolic parameters, including plasma glycemia (mmol/l).
Effect of natural supplement on metabolic parameters including plasma insulinemia and HOMA (homeostatic model assessment) index | Change from baseline to 6 months of the supplementation
  Effect of natural supplement containing chlorogenic acid and luteolin on metabolic parameters, including plasma insulinemia (pmol/L) that with glycemia will be combined to report HOMA index.

SECONDARY OUTCOMES:
Effect of natural supplement on cardio-metabolic parameters including plasma cytokines | Change from baseline to 6 months of the supplementation
  Effect of natural supplement containing chlorogenic acid and luteolin on cardio-metabolic parameters, including plasma cytokines (inflammatory markers and adipokines) (pg/ml), that will be assessed using available enzyme-linked immunosorbent assay (ELISA) kits.
Effect of natural supplement on cardio-metabolic parameters including plasma lipoproteins | Change from baseline to 6 months of the supplementation
  Effect of natural supplement containing chlorogenic acid and luteolin on cardio-metabolic parameters, including atherogenic lipoproteins as well as the analysis of the full spectrum of lipoprotein subclasses by gel electrophoresis.
Effect of natural supplement on cardio-metabolic parameters including subclinical atherosclerosis | Change from baseline to 6 months of the supplementation
  Effect of natural supplement containing chlorogenic acid and luteolin on cardio-metabolic parameters, including subclinical atherosclerosis assessed by carotid intima-media thickness (CIMT) (mm).
Effect of natural supplement on cardio-metabolic parameters including fatty liver index | Change from baseline to 6 months of the supplementation
  Effect of natural supplement containing chlorogenic acid and luteolin on cardio-metabolic parameters, including fatty liver index, a noninvasive method used for steatosis detection and quantification.

CONTACTS AND LOCATIONS:
Overall Officials: Manfredi Rizzo, MD, PhD, Principal Investigator — University Hospital of Palermo, Italy
Locations (1):
- University Hospital of Palermo, Palermo, Palrmo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alberti KG, Eckel RH, Grundy SM, Zimmet PZ, Cleeman JI, Donato KA, Fruchart JC, James WP, Loria CM, Smith SC Jr; International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009 Oct 20;120(16):1640-5. doi: 10.1161/CIRCULATIONAHA.109.192644. Epub 2009 Oct 5. PMID 19805654